CLINICAL TRIAL: NCT05386797
Title: Geniculate Artery Embolization for the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB21-0641
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis
Keywords: Embolization
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geniculate Artery Embolization arm (Experimental)
  Interventions: Procedure: Geniculate Artery Embolization

INTERVENTIONS:
Procedure: Geniculate Artery Embolization — The GAE procedure involves the use of an embolization agent to block blood flow to specific areas of the knee. Under sedo-analgesia, access to the target vessels is gained through the femoral or radial artery. GAE is performed with angiography to visualize blood vessels to assess the affected knee joint and ensure successful treatment.

SUMMARY:
Osteoarthritis (OA) is a highly prevalent degenerative joint disease that contributes to chronic pain and disability in approximately 10% of people over the age of 55. With 25% of Canadians expected to be aged 55 or older by 2036, an increasing number of Canadians will be impacted by knee OA. In affected individuals the risk of medical co-morbidities is increased which can lead to adverse cardiovascular outcomes, depression, and poorer quality of life. Current conservative therapy includes oral analgesia, lifestyle modification, corticosteroid injection, and viscosupplementation. These current conservative measures have variable responses. In patients who would prefer to avoid surgery or are not surgical candidates safe and consistently effective treatment options are lacking.

Geniculate artery embolization (GAE) is a minimally invasive alternative with low risk of complications that has shown promise in exploratory studies. GAE provides benefit by disrupting angiogenesis in the knee which can contribute to chronic inflammation of the affected joint, and helps prevent the growth of new sensory nerve fibers which can reduce the pain associated with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. VAS score of at least 50 mm for knee pain
2. Pain resistant to at least 3 months of conservative therapy (including medical therapy, physiotherapy, intra-articular cortisone or viscosupplement injection).
3. Age > 40 years
4. Radiographs demonstrating knee osteoarthritis on same side as pain
5. Patient not a surgical candidate or declines surgical management

Exclusion Criteria:

1. Radiographically severe knee osteoarthritis (Kellgren-Lawrence grade >2)
2. Severe non-knee related lower limb pain with VAS > 50 mm.
3. Local infection and inflammatory arthritis.
4. Malignancy
5. Previous knee surgery
6. Bleeding risk - known hematologic disease increasing risk of bleeding, pre-procedure INR > 1.4, pre-procedure PTT > 40 seconds or pre-procedure platelets < 50,000/uL
7. Known chronic renal failure or eGFR < 45
8. ECOG grade > 2
9. Patient weight > 300 lbs
10. Patient unreliable for follow up

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | 3 months
  To measure the proportion of patients achieving at least 50% pain reduction by the visual analogue pain score (VAS) after GAE for the treatment of pain due to knee osteoarthritis

SECONDARY OUTCOMES:
Procedure related complications | 30 days
  To measure the incidence of minor and major procedure related adverse events
Pain Reduction | 1 month and 6 months
  To measure the proportion of patients achieving at least 50% pain reduction by the visual analogue pain score (VAS) after GAE for the treatment of pain due to knee osteoarthritis
Pain, stiffness and physical function | 1, 3 and 6 months
  To measure the average improvement in the Western Ontario and McMaster University Osteoarthritis Index (WOMAC) after GAE
Pain medication required | 1, 3, and 6 months
  5. To measure proportion of patients achieving reduction in pain medication required, both in number and dose after GAE

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Hospital, Calgary, Canada